CLINICAL TRIAL: NCT00517985
Title: Duloxetine for Perimenopausal Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F1JUSX026
Record Dates: First submitted 2007-03-09; First posted 2007-08-17 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Major Depressive Disorder
Keywords: perimenopausal depression; duloxetine; cymbalta; major depressive disorder; women
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Duloxetine — During the current study, for a short period of time participants will receive a placebo (a pill that looks like the study drug but which does not contain any medication), although during the majority of the study, participants will be receiving the actual study medication (Duloxetine). The initial dose of Duloxetine to be given will be a 30 mg dose with the dosage increased over time to 60 mg per day. This study will be blinded, meaning that participants will not know whether they are taking placebo or the study drug. However, all subjects will receive duloxetine for the majority of the time they are enrolled in the trial. Investigators will know when subjects are receiving the placebo but in order to maintain the blinding of this study, the study staff will not be able to tell participants when they are taking placebo and when they are taking Duloxetine.

SUMMARY:
Recently, antidepressants have been explored as a class of medications to treat major depression in the context of perimenopause, as well as the somatic symptoms of perimenopause (such as hot flashes). Duloxetine (Cymbalta) is one of the newer antidepressants approved for the treatment of Major Depressive Disorder (MDD). Therefore, the current study is designed to assess the efficacy of duloxetine in a sample of women who are perimenopausal and meet criteria for MDD. We will assess impact on MDD and perimenopausal symptoms.

DETAILED DESCRIPTION:
Over twenty percent of women will experience a major depressive episode in their lifetimes, a prevalence that reflects a greater risk than is found among men. Perimenopausal depression, postpartum depression, and unpleasant, disturbing emotional and physical symptoms that occur just before monthly menstrual periods have been shown to occur during times of fluctuating levels of estrogen and other gonadal hormones.

Perimenopause is commonly defined as a time of hormonal fluctuation that typically occurs in women 40-55 years of age with changes in menstrual patterns. It has been demonstrated that women may be at particularly high risk for depressive symptoms during perimenopause due to declining levels of estrogen. In a previous study, women at risk for postpartum depression were found to benefit from estrogen replacement therapy. However, hormone replacement therapy (HRT) has become increasingly controversial in light of the findings of the Women's Health Initiative study that determined that women who received estrogen plus progestin were slightly more likely to suffer from coronary heart disease, strokes, blood clots in the lungs, and invasive breast cancer. Since the report of these results, HRT use has declined and as an alternative treatment for depression, antidepressants have been increasingly utilized for perimenopausal women. Fluoxetine, paroxetine, and venlafaxine are members of a new class of drugs called selective serotonin reuptake inhibitors (SSRIs) and which have all been demonstrated to be beneficial in the treatment of hot flashes. Recently, a new second-generation drug, Duloxetine (Cymbalta), has also been approved for the treatment of major depression. This drug is a member of a class of compounds that are referred to as serotonin-norepinephrine reuptake inhibitors (SNRIs). The method by which Duloxetine and members of this group achieve their effect is similar to that of the other antidepressant agents that have been used. Recent studies have indicated that Duloxetine appears to provide relief for both the mood and physical components of perimenopause.

In order to continue studying the benefits of Duloxetine in subjects with perimenopause, this study is designed to enroll 20 perimenopausal women with depression in a 9-week trial. Subjects cannot be enrolled in the study if they are currently using hormone replacement therapy and all patients must meet the criteria for a major depressive episode, which will be verified by the standardized protocol for establishing depression, the Structured Clinical Interview for DSM-IV (SCID).

Subjects enrolled in the study, will undergo 7 total clinic visits during a 9-week study period. The first visit will last approximately 3 hours with all other visits taking approximately 45 minutes. During the 1st visit, medical and psychiatric history will be reviewed and blood will be drawn (approximately 3 teaspoons). Blood will be used for routine laboratory testing. Urine will also be collected for a pregnancy test.

For Major Depressive Disorder, the FDA has recommended that a total dose of 40 mg/day (20 mg taken twice a day) to 60 mg/day (given either once a day or as 30 mg twice a day) be administered without regard to meals. While a 120 mg/day dose has been shown to be safe and effective, there is no evidence that doses higher than 60 mg confer additional significant benefit, and the higher dose is clearly less well tolerated. During the current study, for a short period of time participants will receive a placebo (a pill that looks like the study drug but which does not contain any medication), although during the majority of the study, participants will be receiving the actual study medication (Duloxetine). The initial dose of Duloxetine to be given will be a 30 mg dose with the dosage increased over time to 60 mg per day. This study will be blinded, meaning that participants will not know whether they are taking placebo or the study drug. However, all subjects will receive duloxetine for the majority of the time they are enrolled in the trial. Investigators will know when subjects are receiving the placebo but in order to maintain the blinding of this study, the study staff will not be able to tell participants when they are taking placebo and when they are taking Duloxetine.

After the consent forms are read and signed, participants will undergo a Structured Clinical Interview for DSM-IV (SCID) interview. In addition, symptoms will also be rated by rating scales that include the Clinical Global Impression (CGI), the Greene Climacteric Scale (GCS) and the Hamilton Depression Rating Scale (HAM-D (17-item)). To determine functional assessment in all participants, the Global Assessment Scale (GAF) will be used. All participants will also undergo an interview that will include a psychiatric and substance use history (including collection of data regarding the use of alcohol, tobacco, and illicit substances).

Medical screening will occur in conjunction with the initial entry interview. All patients must have had a gynecologic exam within the past year and if not, study personnel will provide a referral for an exam. The investigators will review the patient's medical history. Laboratory tests will include thyroid function tests (TFTs), liver function tests (LFTs), renal panel, pregnancy tests, and complete blood count (CBC). Subjects will also complete the Greene Climacteric Scale, which is used to quantify the severity of perimenopausal symptoms.

At each of the visits, all participants will be administered the CGI, HAM-D, and GCS questionnaires/surveys in addition to The Greene Climacteric Scale, which will be used to quantify symptoms of perimenopause. Also, participants will be asked at each visit if they have missed any doses during that particular week. Each of the office visits will last approximately 45 minutes. If necessary, telephone contact with investigators is permissible and will be available 24 hours/day for emergencies.

Safety and tolerability will be assessed throughout the study. At each study visit, information on any side effects that may have occurred will be collected. In the rare event that a side effect or adverse event does occurs, participants will be able to contact any of the study's research clinicians. Emergency contact personnel will be on-call 24 hours per day, seven days per week.

ELIGIBILITY:
Inclusion Criteria:

* Women age 40 years old or older.
* Perimenopausal symptoms of at least 3 months duration, including irregular periods and/or hot flashes.
* Minimum score of 15 on the Hamilton Rating Scale for Depression (17-item).
* Subjects must be able to be treated on an outpatient basis.
* Subjects must be able to provide written informed consent.

Exclusion Criteria:

* Subjects presently taking antidepressant medication.
* Subjects currently using hormone replacement therapy.
* Subjects who are pregnant.
* Subjects who have hepatic disease.
* Other Axis I disorders, except Generalized Anxiety Disorder or Panic Disorder.
* "Uncontrolled" narrow angle glaucoma.
* Known hypersensitivity to duloxetine or any of the inactive ingredients.
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of study drug administration or potential need to use an MAOI during the study or within 5 days of discontinuation of study drug.
* Presence of psychotic symptoms.
* History of mania or hypomania.
* Hamilton Rating Scale for Depression (HAM-D) suicide item score > 2.
* End stage renal disease or severe renal impairment.
* Abnormal uterine bleeding that has not been evaluated by a gynecologist (heavy or prolonged uterine bleeding, menstrual periods occurring more frequently than every 3 weeks, bleeding after sexual intercourse, spotting between periods).

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Reduction of the initial HAM-D by 50% or more at week 9 of the trial | 9 Weeks
Reduction of the HAM-D score to less than or equal to 7 at week 9 | 9 Weeks
Change of CGI score achievement to "very much improved" or "much improved" at week 9 | 9 Weeks
A 50% decrease in the GCS at week 9. | 9 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathy W Smith, M.D., Principal Investigator — University of Arizona: Department of Psychiatry
Locations (1):
- Women's Mental Health Program; University of Arizona; Department of Psychiatry, Tucson, Arizona, United States